CLINICAL TRIAL: NCT00594243
Title: Feasibility of Mindfulness Meditation for Adults 65+ With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Natalia Morone/Principal Investigator, University of Pittsburfh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0404190
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 8-week mindfulness based stress reduction program
  Interventions: Behavioral: Mindfulness based stress reduction program
- Wait-list control (Active Comparator): Wait-list received no intervention during the time the treatment group received the 8-week program
  Interventions: Other: Wait-list control

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction program — 8-week mindfulness based stress reduction program
  Arms: Intervention
Other: Wait-list control — No treatment given.
  Arms: Wait-list control

SUMMARY:
This pilot feasibility experimental study is designed as a randomized wait-list controlled trial of mindfulness meditation for CLBP. A sample of 37 older adults 65 years of age and older will be recruited from a chronic pain clinic, posted flyers, and newspaper advertisements over a 6-month period. Eligibility will be determined by self-report from a checklist reviewed with potential participants over the phone (see appendix for checklist). Pre-intervention study participants will be consented and study measures obtained. After consent and baseline measures, participants will be randomized in blocks of six using a simple randomization process with no stratification using a table of random numbers. After randomization, participants in the intervention group will receive the intervention of eight weekly 90-minute mindfulness meditation sessions. Instead of waiting until all 37 participants have been recruited into the study to do the intervention, the intervention will be done on a rolling basis. This means there will be a minimum of 6 participants per intervention group, with the possibility of three separate intervention groups. If recruitment goes better than expected, then we will offer the intervention to all 18 participants at one time. Controls will not receive any intervention during this time. Immediately post-intervention the measures will be administered again to participants and wait-list controls. Once the intervention is complete and participants and wait-list controls have completed post-intervention measures the mindfulness meditation program will be offered to the wait-list controls. We will try to combine the wait-list controls into one eight-week program. 3 months after the intervention is completed, participants will be asked to complete the measures a third time and any mindfulness meditation they continue to do at home will be quantified.

The primary hypotheses are:

1. We expect to be able to recruit 37 eligible individuals with CLBP into the study within a six-month period.
2. We expect participants randomized to the mindfulness meditation intervention to meet an adherence standard of attending 75% of the 8 weekly 90-minute sessions.
3. We expect mindfulness meditation will result in a moderate effect size difference (0.5) between the intervention participants and wait-list control participants on outcome measures of pain, mood, physical function, attention, and QOL.

ELIGIBILITY:
Inclusion Criteria:

All participants will be included if they are:

1. 65 years of age or older,
2. have intact cognition (Mini-Mental Status Exam (MMSE) >23),
3. CLBP, defined as moderate pain occurring daily or almost every day for at least the previous three months, and
4. speak English.

Exclusion Criteria:

They will be excluded if they:

1. do not meet the above inclusion criteria,
2. have previously participated in a mindfulness meditation program, and
3. have serious underlying illness (like malignancy, infection, unexplained fever, weight loss or recent trauma) causing their pain.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia E Morone, MD, MSc, Principal Investigator — University of Pittsburgh